CLINICAL TRIAL: NCT06185686
Title: Assessing Radiation Induced Alterations in Resting State Brain Networks in Pediatric Brain Tumor Patients
Brief Title: Radiation Induced Alterations in Resting State Brain Networks in Pediatric Brain Tumor Patients
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); The Foundation for Barnes-Jewish Hospital (Other); Children's Cancer Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: 202312104
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor, Primary
Keywords: Proton therapy; Radiation; Brain tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Brain tumor patients receiving proton radiation therapy: Patients between 8 and 21 years old (inclusive) with a newly diagnosed primary brain tumor that will be treated with proton radiation therapy
  Interventions: Other: Cognitive testing; Device: Resting State MRI/Precision functional mapping

INTERVENTIONS:
Other: Cognitive testing — NIH Toolbox Cognitive Battery and the Novel Cognitive Measure (NCM)
Device: Resting State MRI/Precision functional mapping — At baseline (before the end of radiation therapy) and approximately 12 months after the completion of radiation therapy.
  Other Names: RSFC MRI

SUMMARY:
With modern therapy, the survival rate for pediatric brain tumor patients has significantly improved, with over 70% of patients surviving their disease. However, this progress often comes at the cost of substantial morbidity, with cognitive deficits being the primary obstacle to independent living. Robust predictors of cognitive decline and a comprehensive understanding of the underlying mechanisms of cognitive injury remain elusive. This study will prospectively investigate alterations in brain resting state networks following radiation therapy using functional imaging. The hypothesis is that radiation therapy leads to dose-dependent alterations in functional connectivity in the networks associated with higher level cognition, ultimately leading to cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 and 21 years of age, inclusive
* Newly diagnosed primary brain tumor of any location and any histology that will be treated with proton radiation therapy
* Life expectancy of at least one year
* Able to understand and willing to consent or assent to the research proposed (or that of a legally authorized representative, if applicable), along with consent of legal guardian(s) if applicable

Exclusion Criteria:

* Presence of visual impairment to an extent that the patient is unable to complete the computer testing
* Contraindication to MRI scan (i.e. due to cardiac pacemaker)
* Presence of programmable shunt or dental braces
* Requires sedation for MRI scans

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Treated at Siteman Cancer Center at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Radiation induced effects on functional brain resting state connectivity | Through 1 year follow-up
  The investigators will compare resting state maps of each patient pre- and post-radiation therapy. The investigators will evaluate changes in the resting state architecture and compare to the average results that would be expected from a patient in the same age and sex.
Baseline characteristics of functional network architecture | At baseline (day 1)
  The investigators will assess the unique architecture of brain networks at diagnosis and how significantly this architecture diverges from average healthy controls.
Change in characteristics of functional network architecture | Baseline and 1 year follow-up
  The investigators will assess brain system segregation which is measure of the connection and disconnection between different brain networks. These will be compared within individuals and compared to healthy controls.

SECONDARY OUTCOMES:
Correlation of radiation dose to changes in cognitive performance and resting state network connectivity | At 1 year follow-up
  In an exploratory fashion, the investigators will evaluate the dose of radiation received to each resting state network to determine if functional connectivity changes in a dose dependent manner at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Perkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Saint Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu